CLINICAL TRIAL: NCT05204394
Title: Multicenter, Open-label, Randomized, Active Control Study to Evaluate Efficacy and Safety of Switching to VM-1500A-LAI + 2NRTIs From the 1st Line Standard of Care Therapy
Brief Title: Study to Evaluate Efficacy and Safety of Switching to VM-1500A-LAI + 2NRTIs From the 1st Line Standard of Care Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500ALAI-03
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: HIV-1-infection
Keywords: HIV-1; LAI
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VM-1500A-LAI 600mg (Experimental): 20mg Elpida® 2 weeks run-in period followed by VM-1500A-LAI 600mg i / m Q4W injections with the background of oral 2NRTIs QD.
  Interventions: Drug: VM-1500A-LAI
- VM-1500A-LAI 900mg (Experimental): 20mg Elpida® 2 weeks run-in period followed by VM-1500A-LAI 900mg i / m Q4W injections with the background of oral 2NRTIs QD.
  Interventions: Drug: VM-1500A-LAI
- Standard or Care (Other): Any approved 1st line oral HIV treatment regimen
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: VM-1500A-LAI — Injectable nanoformulation of depulfavirine (parent drug of elsulfavirine)
  Other Names: VM-1500A; Depulfavirine
  Arms: VM-1500A-LAI 600mg; VM-1500A-LAI 900mg
Other: Standard of Care — Any oral 1st line approved HIV treatment regimen
  Other Names: SoC
  Arms: Standard or Care

SUMMARY:
Multicenter, open-label, randomized, active control study to evaluate efficacy and safety of switching to VM-1500A-LAI + 2NRTIs from the 1st line standard of care therapy for 48 weeks. The 1st part of the study will select one of 2 dose cohorts: 600mg or 900mg.

DETAILED DESCRIPTION:
Eligible patients will be randomized (1:1:1) into 3 treatment groups - LAI 600 (ELPIDA+VM-1500A-LAI 600 mg), LAI 900 (ELPIDA+VM-1500A-LAI 900 mg), and Standard of Care (SoC) therapy. Patients of LAI groups will be assigned by ELPIDA®, 20 mg capsules (and same 2NRTIs) daily therapy for 4 weeks, then one IM injection of 1200 mg VM-1500A-LAI followed by 5 IM monthly injections of 600 mg or 900 mg VM-1500A-LAI QM. When all patients in the VM-1500A-LAI 600mg and VM-1500A-LAI 900 mg dose cohorts complete 24 weeks, the interim analysis will be performed in order to select the dosage regimen for VM-1500A-LAI to continue for additional 28 weeks for a total of 52 weeks of treatment. The analysis will be based on efficacy assessment (number of patients treated with VM1500-LAI who showed the viral load ≥ 50 copies/ml at Week 24 using FDA snapshot algorithm as well as on the basis of a safety and tolerability assessment (assessment of the frequency and severity of AEs associated with the study drug). The optimal dosage regimen will be selected by the IDMC.

4 weeks after the End of Treatment visit, subjects will come for the Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information Sheet and Informed Consent Form
2. Men and women aged 18 or older at the time of signing the informed consent;
3. HIV-1 infection confirmed serologically by ELISA or immunoblot analysis (or documented HIV-1 infection);
4. Stable doses of standard-of-care antiretroviral therapy (NNRTI + 2NRTI) for at least 6 months prior screening;
5. Serological confirmation of adequate virological suppression within 6 and 12 months before screening as documented by :

   * HIV-1 RNA plasma level < 50 copies/ml at screening;
   * СD4+ Т-cells count ≥ 200 cells/mm3 at screening;
6. Adequate organ function as documented by laboratory test results;
7. Female patients must be postmenopausal not less than 2 years, surgically sterile, or if of child-bearing potential, must use two reliable forms of contraception from screening to 3 months after the end of dosing; two reliable forms of contraception include use of condom with spermicide by male partner, or diaphragm with spermicide, or condom use by male partner and diaphragm, or condom use by male partner and non-hormonal intrauterine device.
8. Male patients must use two reliable forms of contraception from screening to 3 months after the end of dosing; two reliable forms of contraception include condom with spermicide, or diaphragm use by female partner with spermicide, or condom and diaphragm use by female partner, or condom and intrauterine device use by female partner.

Exclusion Criteria:

1. Acute hepatitis or cirrhosis of the liver of any etiology; HBsAg or antibodies to hepatitis C (in the case of Anti-HCV +, the exclusion criterion must be confirmed by determining a positive HCV RNA test) at screening;
2. Signs of acute infection or presence of syphilis, hepatitis A, Toxoplasma gondii, cytomegalovirus, gonorrhea and Chlamydia trachomatis tests results within 30 days prior to screening
3. Patients with known or suspected active Coronavirus Disease 2019 (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment (World Health Organization [WHO] definitions).
4. Opportunistic infections referred to Category C of the classification of the Center for disease control (CDC), dated 2008, except for Kaposi's sarcoma not requiring system therapy (Appendix 2)
5. History of tuberculosis of any localization or ongoing at screening according to chest x-ray (in frontal and lateral projections) and other serology testing;
6. History of malignant neoplasms (except for basal cell epithelioma or squamous cell carcinoma of skin and in situ cervical carcinoma, which were resected and healed more than 5 years ago);
7. Participation in other clinical studies or therapy with other study drugs within 3 months or 5 half-lives before Screening, whichever is longer.;
8. Treatment with immunomodulators (interferons, interleukins), immune-suppressive therapy (cyclosporins), glucocorticoids 1 month before screening

   a. Washout from these medications for the purpose of participation in tis clinical trials needs to be done safely and only if medically acceptable.
9. Current alcoholic or drug addiction, which the researcher may think to hinder the patient to take part in the study and adhere to all requirements per protocol
10. Hypersensitivity to any component of the study drug such as hypersensitivity to lactose intolerance, or the presence of contraindications to the appointment of ELPIDA® or ART drugs;
11. Treatment with prohibited drugs from the list of "prohibited drugs" (Appendix 3);
12. Signs of manifest uncontrolled and/or unstable concomitant disease, e.g., disorders of nervous, respiratory, systems, kidneys, liver, endocrine system and gastrointestinal tract, which as the Investigator may think could prevent the patient from participation in the study;
13. Clinically significant cardiovascular diseases including:

    * Myocardial infarction within 12 months before screening
    * Unstable angina within 12 months before screening
    * Congestive heart failure Class III or IV according to the New York Heart Association criteria (NYHA)
    * Clinically significant ventricular arrhythmia including ventricular tachycardia, ventricular fibrillation, history of cardiac arrest, atrioventricular block (Mobitz II or III), use of cardiostimulator
    * QTc interval > 450 ms in men or 470 ms in women (ECG) (calculated according to Fredericia formula), or a diagnosis of long QT syndrome
    * Hypotension (systolic blood pressure < 86 mm Hg or bradycardia with a heart rate of < 50 beats per minute (ECG) except when caused by medications (e.g. beta-blockers).

      * Uncontrolled/unstabe arterial hypertension (systolic arterial pressure > 170 millimeters of mercury or diastolic blood pressure > 105 millimeters of mercury)
14. Systemic autoimmune disorders and connective tissue diseases, which require prior or current treatment with systemic glucocorticoid drugs, cytostatics or penicillamine;
15. Pregnant or lactating women or women planning to get pregnant during the clinical study;
16. The patient has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
17. History of hypersensitivity (analphylaxis) reactions upon intramuscular injection
18. Positive breath alcohol test or/and positive urine drug screen
19. Inability to read or write; unwillingness to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator believes may affect the study results or subject's safety and prevent the subject from further participation in the study; any other concomitant medical or serious psychological conditions making the subject not eligible to participate in the clinical study restrict the legality of obtaining the Informed Consent or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with plasma HIV-1 RNA level > 50 copies/mL | 48 Weeks
  Proportion of participants with plasma HIV-1 RNA level > 50 copies/mL at Week 48 using the snapshot algorithm (FDA).

SECONDARY OUTCOMES:
Percentage of patients with undetectable viral load | 48 Weeks
  Percentage of patients with HIV-1 RNA < 50 copies/ml at Week 48
Proportion of patients with Confirmed Virologic Failure | 48 Weeks
  Proportion of patients with Confirmed Virologic Failure (two consecutive plasma HIV-1 RNA levels > 200cmL after prior suppression to < 200copies/ml) at Week 48
Change in the absolute lymphocyte counts | 48 Weeks
  Change in the absolute CD4+ and CD8+ lymphocyte counts over 48 weeks
Percentage of patients with developed HIV-1 resistance | 48 Weeks
  Percentage of patients who develop HIV-1 resistance to study therapy over 48 weeks
Incidence of AEs / SAEs | 48 Weeks
VM-1500A plasma concentration | 48 Weeks
  To assess PK parameters of VM-1500A-LAI

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Pokrovskaya, PhD, Principal Investigator — Central Research Institute of Epidemiology of Rospotrebnadzor
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution of the Central Research Institute of Epidemiology of Rospotrebnadzor, Moscow
  - St. Petersburg State Medical Institution " Center for AIDS and Infectious Diseases", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No